CLINICAL TRIAL: NCT03698149
Title: A High-Performance ECoG-based Neural Interface for Communication and Neuroprosthetic Control
Brief Title: ECoG BMI for Motor and Speech Control
Acronym: BRAVO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karunesh Ganguly (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Karunesh Ganguly, Associate Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 17-23028; U01DC018671 (NIH)
Record Dates: First submitted 2018-08-21; First posted 2018-10-05 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: ALS; SCI - Spinal Cord Injury; Stroke; Multiple Sclerosis; Muscular Dystrophies
MeSH Terms: conditions — Spinal Cord Injuries; Stroke; Multiple Sclerosis; Muscular Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Electrocorticography-based brain computer interface (Experimental)
  Interventions: Device: PMT/Blackrock Combination Device

INTERVENTIONS:
Device: PMT/Blackrock Combination Device — PMT Subdural Cortical Electrodes/Blackrock NeuroPort Array and NeuroPort System

SUMMARY:
Test the feasibility of using electrocorticography (ECoG) signals to control complex devices for motor and speech control in adults severely affected by neurological disorders.

DETAILED DESCRIPTION:
ECoG is a type of electrophysiological monitoring that uses electrodes placed directly on the exposed surface of the brain to record electrical activity. With this ECoG-based neural interface, study patients will undergo training and assessment of their ability to control a complex robotic system and to determine if ECoG brain signals can be used to produce speech.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 21
2. Limited ability to use upper limbs, based on neurological examination, due to stroke, amyotrophic lateral sclerosis (ALS), multiple sclerosis, cervical spinal cord injury, brainstem stroke, muscular dystrophy, myopathy or severe neuropathy.
3. Disability, defined by a 4 or greater score on the Modified Rankin Scale, must be severe enough to cause loss of independence and inability to perform activities of daily living.
4. If stroke or spinal cord injury, at least 1 year has passed since onset of symptoms
5. Must live within a two-hour drive of UCSF

Exclusion Criteria:

1. Pregnancy or breastfeeding
2. Inability to understand and/or read English
3. Inability to give consent
4. Dementia, based on history, physical exam, and MMSE
5. Active depression (BDI > 20) or other psychiatric illness (active general anxiety disorder, schizophrenia, bipolar disorder, obsessive-compulsive disorder (OCD), or personality disorders (e.g. multiple personality disorder, borderline personality disorder, etc.)
6. History of suicide attempt or suicidal ideation
7. History of substance abuse
8. Co-morbidities including ongoing anticoagulation, uncontrolled hypertension, cancer, or major organ system failure
9. Inability to comply with study follow-up visits
10. Any prior intracranial surgery
11. History of seizures
12. Immunocompromised
13. Has an active infection
14. Has a CSF drainage system or an active CSF leak
15. Requires diathermy, electroconvulsive therapy (ECT), or transcranial magnetic stimulation (TMS) to treat a chronic condition
16. Has an implanted electronic device such as a neurostimulator, cardiac pacemaker/defibrillator or medication pump, or presence of any head or neck metallic foreign bodies
17. Allergies or known hypersensitivity to materials in the Blackrock NeuroPort Array (i.e. silicone, titanium) or the PMT Subdural Cortical Electrode (silicone, platinum iridium, nichrome)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2018-11-09 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2030-08-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 6 years post-implant period
  The primary endpoint of this study is to determine the incidence of treatment-emergent adverse events associated with the ECoG-based interface
NIDCD Primary Objective 1 | Up to 6 years post-implant period
  To enable communication via text decoded from neural signals.
NIDCD Primary Objective 2 | Up to 6 years post-implant period
  To enable communication via synthesized speech decoded from neural signals.

SECONDARY OUTCOMES:
NIDCD Secondary Objective 1 | Up to 6 years post-implant period
  To evaluate communication via text decoded from neural signals.
NIDCD Secondary Objective 2 | Up to 6 years post-implant period
  To evaluate communication via synthesized speech decoded from neural signals.

CONTACTS AND LOCATIONS:
Overall Officials: Karunesh Ganguly, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silva AB, Liu JR, Anderson VR, Kurtz-Miott CM, Hallinan IP, Littlejohn KT, Brosler SC, Tu-Chan A, Ganguly K, Moses DA, Chang EF. Implications of shared motor and perceptual activations on the sensorimotor cortex for neuroprosthetic decoding. J Neural Eng. 2025 Aug 7;22(4):046039. doi: 10.1088/1741-2552/adf50e. PMID 40720979
- [Derived] Shah AM. Unlocking Naturalistic Speech With Brain-Computer Interface. Artif Organs. 2025 Jul;49(7):1087-1088. doi: 10.1111/aor.15021. Epub 2025 May 12. PMID 40353311
- [Derived] Silva AB, Liu JR, Anderson VR, Kurtz-Miott CM, Hallinan IP, Littlejohn KT, Brosler S, Tu-Chan A, Ganguly K, Moses DA, Chang EF. Implications of shared motor and perceptual activations on the sensorimotor cortex for neuroprosthetic decoding. medRxiv [Preprint]. 2025 Apr 28:2025.04.24.25326368. doi: 10.1101/2025.04.24.25326368. PMID 40343020
- [Derived] Metzger SL, Liu JR, Moses DA, Dougherty ME, Seaton MP, Littlejohn KT, Chartier J, Anumanchipalli GK, Tu-Chan A, Ganguly K, Chang EF. Generalizable spelling using a speech neuroprosthesis in an individual with severe limb and vocal paralysis. Nat Commun. 2022 Nov 8;13(1):6510. doi: 10.1038/s41467-022-33611-3. PMID 36347863
- [Derived] Moses DA, Metzger SL, Liu JR, Anumanchipalli GK, Makin JG, Sun PF, Chartier J, Dougherty ME, Liu PM, Abrams GM, Tu-Chan A, Ganguly K, Chang EF. Neuroprosthesis for Decoding Speech in a Paralyzed Person with Anarthria. N Engl J Med. 2021 Jul 15;385(3):217-227. doi: 10.1056/NEJMoa2027540. PMID 34260835